CLINICAL TRIAL: NCT02244684
Title: Effects of Maternal Folate and Folic Acid Supplementation on DNA Methylation in the Newborn Infant
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Young In Kim, Senior Scientist, Unity Health Toronto
Other Study IDs: 10-246
Record Dates: First submitted 2014-09-02; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Pregnancy; Maternal Nutrition; Fetal Health; Epigenetics; Maternal B Vitamins
Keywords: Folate; Folic Acid; One-Carbon Nutrients; Epigenetics; Pregnancy; Fetal Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pregnant women

SUMMARY:
An overwhelming body of evidence of the protective effect of folic acid supplementation on neural tube defect affected pregnancies led to mandatory folic acid fortification in Canada in 1998. Folate is an important co-factor in the transfer of one-carbon units essential in DNA synthesis, repair, and methylation reactions, aberrations of which have been implicated in the pathogenesis of several chronic diseases including cancer. Epigenetic reprogramming occurs in utero and has the potential to be modulated by the methyl donor supply of which folate is a contributor. Animal studies have shown maternal folate exposure can modulate epigenetic changes in the offspring, however, there is limited evidence of this relationship in humans. The aim of this research is to determine the effects of maternal dietary folate and supplemental folic acid intake during the periconceptional and in utero periods on global and gene-specific DNA methylation in human infants. This is a prospective observational study involving 368 Canadian mother-child pairs recruited from St. Michael's Hospital in Toronto, Ontario. Dietary and demographical information was collected from consenting pregnant women at study baseline (12-16 weeks gestation) and in the third trimester (34-37 weeks gestation). Maternal blood samples were obtained at baseline and prior to delivery and a sample of umbilical cord blood was collected at parturition to measure levels of folate status. Global and gene-specific DNA methylation in umbilical cord blood will be correlated with cord and maternal folate status. The data will be analyzed using separate ordinary least squares (OLS) regressions. Results from this study will contribute to a better understanding of how maternal folate and folic acid intake can modulate epigenetic modifications in the offspring and potentially have an effect on disease susceptibility later in life.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy

Exclusion Criteria:

* celiac disease
* Crohn's disease
* irritable bowel disease (IBD)
* gastric bypass surgery
* use of antifolate medications
* banking umbilical cord blood

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women were recruited from obstetrics clinics at St Michael's Hospital, a tertiary teaching hospital affiliated with the University of Toronto.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2010-09; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Global CpG DNA methylation in umbilical cord blood lymphocytes determined by LC/MS-MS | Day 1
  Maternal dietary intake and supplemental use and blood levels of folate/folic acid and other one carbon nutrients in early and late pregnancy will be correlated with global CpG DNA methylation in umbilical cord blood lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Young-In Kim, MD, Principal Investigator — Unity Health Toronto; Deborah O'Connor, RD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Plumptre L, Tammen SA, Sohn KJ, Masih SP, Visentin CE, Aufreiter S, Malysheva O, Schroder TH, Ly A, Berger H, Croxford R, Lamers Y, Caudill MA, Choi SW, O'Connor DL, Kim YI. Maternal and Cord Blood Folate Concentrations Are Inversely Associated with Fetal DNA Hydroxymethylation, but Not DNA Methylation, in a Cohort of Pregnant Canadian Women. J Nutr. 2020 Feb 1;150(2):202-211. doi: 10.1093/jn/nxz232. PMID 31562504
- [Derived] Visentin CE, Masih SP, Plumptre L, Schroder TH, Sohn KJ, Ly A, Lausman AY, Berger H, Croxford R, Lamers Y, Kim YI, O'Connor DL. Low Serum Vitamin B-12 Concentrations Are Prevalent in a Cohort of Pregnant Canadian Women. J Nutr. 2016 May;146(5):1035-42. doi: 10.3945/jn.115.226845. Epub 2016 Apr 13. PMID 27075906
- [Derived] Plumptre L, Masih SP, Ly A, Aufreiter S, Sohn KJ, Croxford R, Lausman AY, Berger H, O'Connor DL, Kim YI. High concentrations of folate and unmetabolized folic acid in a cohort of pregnant Canadian women and umbilical cord blood. Am J Clin Nutr. 2015 Oct;102(4):848-57. doi: 10.3945/ajcn.115.110783. Epub 2015 Aug 12. PMID 26269367
- [Derived] Masih SP, Plumptre L, Ly A, Berger H, Lausman AY, Croxford R, Kim YI, O'Connor DL. Pregnant Canadian Women Achieve Recommended Intakes of One-Carbon Nutrients through Prenatal Supplementation but the Supplement Composition, Including Choline, Requires Reconsideration. J Nutr. 2015 Aug;145(8):1824-34. doi: 10.3945/jn.115.211300. Epub 2015 Jun 10. PMID 26063067
- [Derived] Visentin CE, Masih S, Plumptre L, Malysheva O, Nielsen DE, Sohn KJ, Ly A, Lausman AY, Berger H, Croxford R, El-Sohemy A, Caudill MA, O'Connor DL, Kim YI. Maternal Choline Status, but Not Fetal Genotype, Influences Cord Plasma Choline Metabolite Concentrations. J Nutr. 2015 Jul;145(7):1491-7. doi: 10.3945/jn.115.211136. Epub 2015 May 13. PMID 25972528